CLINICAL TRIAL: NCT05639582
Title: Evaluation of Trabecular Bone Changes in Individuals With Periodontal Disease Using Fractal Analysis
Brief Title: Fractal Analysis Method in Periodontal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Ummuhan Tekin Atay, Principal Investigator, Necmettin Erbakan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Ummuhantekinatay
Record Dates: First submitted 2022-11-26; First posted 2022-12-06 (Actual); Last update posted 2022-12-08 (Actual); Status verified 2022-12

CONDITIONS: Periodontal Diseases
Keywords: Digital Radiography; Fractal Analysis; Periodontitis
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- periodontally healthy individuals (Experimental): 50 subject without any periodontal disease
  Interventions: Other: fractal analysis
- Stage 1 periodontitis (Experimental): 50 subject diagnosed with stage 1 in the periodontal disease classification
  Interventions: Other: fractal analysis
- Stage 2 periodontitis (Experimental): 50 subject diagnosed with stage 2 in the periodontal disease classification
  Interventions: Other: fractal analysis
- Stage 3 periodontitis (Experimental): 50 subject diagnosed with stage 3 in the periodontal disease classification
  Interventions: Other: fractal analysis

INTERVENTIONS:
Other: fractal analysis — fractal analysis is a method that numerically expresses bone changes.

SUMMARY:
In this study, the effects of periodontal disease on alveolar bone were investigated using fractal analysis method.

DETAILED DESCRIPTION:
Background: It is very difficult to objectively evaluate the negative changes in bone structure due to periodontitis. The present study was aimed to evaluate the trabecular bone changes between healthy individuals and periodontitis patients by fractal dimension analysis on digital panoramic radiographs.

Method: The study included 50 periodontally healthy individuals (control group), 50 individuals with Stage 1 periodontitis (S1-P group), 50 individuals with Stage 2 periodontitis (S2-P), and 50 individuals with Stage 3 periodontitis (S3-P), a total of 200 individuals were included. The fractal dimension (FD) value of the trabecular bone in the interproximal space between mandibular first molar and second premolar tooth roots was evaluated using Image J program. The mean fractal dimension values of the two regions were calculated by box counting method.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* Getting a diagnosis of stage 1,2 and 3 periodontitis
* Be diagnosed as periodontally healthy
* Have no barriers to obtaining radiographs
* Not having any systemic disease that may affect periodontal status
* Not smoking and alcohol use
* Volunteer to participate in the study

Exclusion Criteria:

* Those who use drugs that can affect bone metabolism
* Radiographs with poor diagnostic quality
* Root canal treatment or teeth with periapical lesions in the area of interest
* Individuals who have suffered a fracture or trauma that affects the anatomy or integrity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-05-05 (Actual); Study Completion 2021-11-05 (Actual)

PRIMARY OUTCOMES:
Evaluation of the effect of periodontal disease on alveolar bone by fractal analysis | baseline
  Fractal dimension evaluation can give an objective result about the effect of periodontal disease on alveoler bone, since it shows changes in bone trabeculation numerically.

SECONDARY OUTCOMES:
Probing pocket depth | baseline
  Probing pocket depth(PPD) was measured for determining the severity of the disease and clinical outcome. High probing pocket depth shows more severe periodontal disease.
gingival index | baseline
  The differences in gingival index scores between periodontally healthy and periodontitis.The gingival index was recorded for determining and classifying gingival status. The Gingival İndex(GI) scores each site on a 0 to 3 scale with 0 being normal and 3 being severe inflammation characterized by edema, redness, swelling and spontaneous bleeding.
plaque index | baseline
  The differences in plaque index scores between periodontally healthy and periodontitis. Plaque index(PI) was recorded for determining and classifying oral hygiene status. The plaque index(PI) scores each site on a 0 to 3 scale with 0 being no plaque in the gingival area and 3 abundance of soft matter within the gingival pocket and/or on the gingival margin and adjacent tooth surface.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No